CLINICAL TRIAL: NCT05683639
Title: Randomized Clinical Trial in Women Submitted to in Vitro Fertilization: Warming Versus Not Warming of the Follicular Aspiration Needle.
Brief Title: Heated and Non Heated Ovarian Aspiration Needle Protocol
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Collaborators: Guedes da Luz Médicos Associados Sociedade Simples LTDA (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: 60504522.7.0000.5327
Record Dates: First submitted 2022-12-22; First posted 2023-01-13 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2024-03

CONDITIONS: Infertility, Female
MeSH Terms: conditions — Infertility, Female

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard protocol (No Intervention): The standard protocol comprises no heating of the aspiration needle.
- Warming protocol (Experimental): The aspiration needle will be warm-up overnight the day before the oocyte pick-up procedure
  Interventions: Other: warming of the follicular aspiration needle

INTERVENTIONS:
Other: warming of the follicular aspiration needle — the follicular aspiration needle will be heated overnight before the ovarian aspiration procedure.
  Arms: Warming protocol

SUMMARY:
The success of IVF is influenced by factors as cause of infertility and age. Furthermore, there is a large influence of external factors, from the laboratory environment, handling and cultivation of gametes and embryos. The existence of factors capable of affecting the success of the treatment lead to the need of a quality control to attenuate the unfavorable effects.

After ovarian stimulation, follicular aspiration is performed. At this moment, factors such as aspiration technique, needle type and temperature are the main variables to be controlled. It is known that oocytes are the more sensitive cells to temperature fluctuations. Currently, the standard protocol for follicular aspiration does not include the warming of the aspiration needle. However, due to the existing evidence in the literature, that the follicular fluid temperature drops during the aspiration procedure, this work aims to evaluate the influence of a pre warming of the aspiration needle as a new protocol.

DETAILED DESCRIPTION:
The estimated sample was 600 oocytes for each group, totaling a minimum of 1200 oocytes, considering a fertilization rate of 65% in the control group and 73% in the study group, for a power of 80% and p alpha 5%, i.e. , an increase of more than 10% between groups. As there is no data in the literature, when the investigators have this sample an interim analysis to evaluate the data will be performed. The investigators consider 10% a reasonable difference that can (with this sample size) increase by 48 embryos and a possible increase of 7 pregnancies within this sample. Bearing in mind that the average number of oocytes retrieved per patient is 6 oocytes, the investigators estimate that 200 patients will be needed to reach the calculated sample number.

The warm-up protocol will be applied by the embryologists, which consists of heating the follicular aspiration needle to 37 Celsius, overnight, the day before the day of the ovarian aspiration procedure.

The variables that will be compared between the studied groups are the rates of oocyte retrieval, maturity (MII), fracture, atresia, fertilization rates and discarded embryos.

Continuous variables will be analyzed using Student's t test if they have normal distribution, for comparison of means between two independent groups or the Wilcoxon-Mann-Whitney U test if not parametric. Differences between groups will be considered significant when p<0.05.

ELIGIBILITY:
Inclusion Criteria:

* All women submitted to IVF cycles

Exclusion Criteria:

* Women submitted to follicular aspiration due to oocyte cryopreservation
* Patients without oocyte retrieved
* Patients without mature oocyte retrieved
* Procedures with needle replacement

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 179 (Actual)
Dates: Start 2023-01-02 (Actual); Primary Completion 2023-03-01 (Actual); Study Completion 2023-06-01 (Actual)

PRIMARY OUTCOMES:
normal fertilization rate | 16 to 18 hours after fertilization procedure
  Fertilization will be confirmed through the visualization of the presence of two pronuclei

SECONDARY OUTCOMES:
number of oocyte retrieved | immediately after ovarian aspiration procedure
  the total number of oocytes captured in the ovarian aspiration procedure
number of mature oocyte | 3 hours post ovarian aspiration
  total number of MII
oocyte damage rate | 3 hours post ovarian aspiration
  the number of fractured oocytes or atresia
abnormal fertilization rate | 16 to 18 hours after fertilization procedure
  the total number of zygotes with three or more pronuclei

CONTACTS AND LOCATIONS:
Overall Officials: João da Cunha Filho, PhD, Study Director — Hospital de Clínicas de Porto Alegre
Locations (1):
- Insemine Human Reproduction Centre, Porto Alegre, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: No